CLINICAL TRIAL: NCT01387906
Title: Latisse(Bimatoprost .03% Opthalmic Solution) for the Treatment of Hypotrichosis of the Eyebrows: Latisse Versus Placebo
Brief Title: Latisse (Bimatoprost .03% Opthalmic Solution) for the Treatment of Hypotrichosis of the Eyebrows: Latisse Versus Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kenneth Beer (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Kenneth Beer, Investigator, Beer, Kenneth R., M.D., PA
Organization: Beer, Kenneth R., M.D., PA (Individual)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Latisse2010
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Hypotrichosis
Keywords: mild; moderate
MeSH Terms: conditions — Hypotrichosis; Lymphoma, Follicular | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical bimatoprost for eyebrows (Experimental): Topical bimatoprost will be applied to areas of the eyebrow that have diminished eyebrows (hypotrichosis).
  Interventions: Drug: topical bimatoprost

INTERVENTIONS:
Drug: topical bimatoprost — topical bimatoprost will be applied one drop to each eyebrow each night.
  Other Names: bimatoprost, Latisse, eyebrows

SUMMARY:
The primary purpose of this study is to assess efficacy and safety of Latisse (bimatoprost .03% ophthalmic solution) applied to the lateral and medial eyebrows. The primary outcome is a increase in overall eyebrow prominence as measured by at least a 1-grade increase on the Global Eyebrow Assessment (GEyA) scale, from baseline to the end of the treatment which will be day 270 period.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, female/male subjects of any race, 18-75 years of age.
* Subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study
* Patients with hypotrichosis (thinning) of the eyebrows with a GEyA score of 1 or 2.
* Patient agrees to abstain from any treatment to the eyebrows including: waxing, plucking, threading, laser hair removal, and/or bleaching (excluding the glabella region).
* Able to understand the requirements of the study and sign Informed Consent/HIPAA Authorization forms.
* Written informed consent and written authorization for use or release of health and research information obtained.
* Willing to complete all required study visits, procedures, and evaluations including photography.

Exclusion Criteria:

* Subjects who are pregnant (positive urine pregnancy test), planning to become pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
* Patients with any uncontrolled systemic disease
* Patient with any known disease or abnormality of the eyebrows including eczema and seborrheic dermatitis
* Patients with known or suspected trichotillomania disorder
* Patients with a history of glaucoma and/or increased ocular pressure
* Patients who are currently using an IOP-lowering prostaglandin analog (including Lumigan)
* Patients with a known hypersensitivity to bimatoprost or any other ingredient in Latisse
* Previous cosmetic surgery to the upper face (e.g., periorbital surgery, brow lift, eyelid or eyebrow surgery, etc.).
* Patients with permanent eye and/or eyebrow make-up
* Any eyebrow tint or dye applications within 2 months prior to study entry
* Any planned facial cosmetic procedure that would interfere with the evaluation of the eyebrows
* Participation in another investigational drug or device study within the last 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of Latisse applied to the lateral and medial eyebrow | 10 months
  Increase in overall eyebrow prominence as measured by at least a 1-grade increase on the Global Eyebrow Assessment (GEyA) scale, from baseline to the end of the treatment which will be day 270 period.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Beer, M.D., Principal Investigator — Beer, Kenneth R., M.D., PA
Locations (1):
- Kenneth R. Beer, M.D. ,PA, West Palm Beach, Florida, United States

REFERENCES:
- [Background] Law SK. Bimatoprost in the treatment of eyelash hypotrichosis. Clin Ophthalmol. 2010 Apr 26;4:349-58. doi: 10.2147/opth.s6480. PMID 20463804
- [Background] Bimatoprost 0.03% solution (latisse) for eyelash enhancement. Med Lett Drugs Ther. 2009 Jun 1;51(1313):43-4. No abstract available. PMID 19478690
- See also: eyebrows, bimatoprost, hypotrichosis — http://www.palmbeachcosmetic.com